CLINICAL TRIAL: NCT06539390
Title: Impact of Sedation on Patient Satisfaction, Radiation Exposure, and Complications in Lumbar Transforaminal Epidural Steroid Injections: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Sedation in epidural injection
Record Dates: First submitted 2024-04-24; First posted 2024-08-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pain, Chronic
Keywords: Transforaminal Epidural Injections, Sedation,Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Is Sedation Necessary for Transforaminal Epidural Injections
  Interventions: Other: Transforaminal Epidural Injections?

INTERVENTIONS:
Other: Transforaminal Epidural Injections? — Pain, lumbar disc herniation,Transforaminal Epidural Injections?
  Other Names: Is Sedation Necessary for Transforaminal Epidural Injections?

SUMMARY:
Radicular low back pain due to disc herniation is frequently observed. There are rest, medical treatments, physical medicine modalities, interventional procedures for pain and surgical options in the treatment of lumbar disc herniations. Epidural interventional methods can be applied safely and effectively in patients who do not respond to conservative treatment. Transforaminal epidural steroid injections (TFESE) are frequently used in the interventional treatment of lumbosacral radicular low back pain. TFESE is applied targetedly under fluoroscopy guidance in disc herniation. Therefore, the chance of success increasesTFESE, which is considered a minimally invasive procedure today, is frequently preferred in interventional pain treatments. TFESE can be performed with or without sedation, depending on the preference of the physician and the patient, the patient's comorbidities, the infrastructure of the hospital and the health presentation. There are conflicting and limited studies on whether sedation is necessary in interventional pain procedures.

DETAILED DESCRIPTION:
The study will be conducted by retrospectively scanning the files of patients with paracentral/subarticular protruded disc herniation and who underwent transforaminal epidural steroid injection (TFESE) to the lumbosacral region, at the Algology Department of Kanuni Sultan Süleyman Training and Research Hospital, between January 2021 and January 2024. In order to prevent heterogeneity, magnetic resonance imaging (MRI) of the patients will be evaluated in consultation with a radiologist. will be used. . 201 patients aged 18-65 years, classified as American Society of Anesthesiologists (ASA) 1-3, who underwent unilateral L-TFESI, were included in the study. The patient selection process is shown in Figure 1. The patients' magnetic resonance (MR) images were evaluated by a radiologist with 10 years of experience in the musculoskeletal system. The classification system used in the studies by Pfirmann et al. and Ghahreman et al. was used to grade nerve root compression based on MR imaging. According to this classification system, DH compression was graded as low-grade (1-2) or high-grade (3-4) nerve root compression The Numeric Rating Scale-11 (NRS-11) and Likert scale were recorded on the 4th day and 4th week before and after the procedure. It is stated that the outcome of epidural steroid injections can be predicted from the 4th day onwards

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-65, American Society of Anesthesiologists (ASA) 1-3, who underwent unilateral, single-level TFESE were included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exclusion Criteria:
  * Patients with ASA 4 and above,
  * patients with a history of lumbar surgery,
  * patients with multi-level disc herniation,
  * malignancy,
  * psychosis,
  * patients without MRI imaging,
  * patients with known allergies to the drugs used,
  * patients with bleeding disorders,
  * patients with infection at the injection site, and pregnant patients were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale-11 (NRS-11) | one month
  It is an 11-point numerical scale where patients can rate their pain on a scale of 0 (no pain) to 10 (the most severe pain they have ever felt).

SECONDARY OUTCOMES:
Likert scale | four days
  It is a satisfaction rating scale where satisfaction is rated on a scale of 1 to 5, with 1 being not satisfied at all and 5 being very satisfied, and the higher the score, the higher the satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided